CLINICAL TRIAL: NCT02785952
Title: A Phase III Randomized Study of Nivolumab Plus Ipilimumab Versus Nivolumab for Previously Treated Patients With Stage IV Squamous Cell Lung Cancer and No Matching Biomarker (Lung-Map Sub-Study)
Brief Title: Lung-MAP: Nivolumab With or Without Ipilimumab as Second-Line Therapy in Treating Patients With Recurrent Stage IV Squamous Cell Lung Cancer and No Matching Biomarkers
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1400I; NCI-2016-00050 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1400I; S1400I (Other: SWOG); S1400I (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Results first posted 2022-01-11 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Squamous Cell Lung Carcinoma; Stage IV Squamous Cell Lung Carcinoma AJCC v7
MeSH Terms: interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 and ipilimumab IV over 60 minutes on day 1 of every third course (every 42 days). Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (nivolumab) (Active Comparator): Patients receive nivolumab IV over 30 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm I (nivolumab, ipilimumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase III trial compares nivolumab with ipilimumab and nivolumab alone in treating patients with stage IV squamous cell lung cancer that has come back after previous treatment. This is a "non-match" sub-study that includes all screened patients not eligible for a biomarker-driven sub-study. Monoclonal antibodies, such as nivolumab and ipilimumab, may be able to shrink tumors. It is not yet known whether nivolumab works better with or without ipilimumab in treating patients with squamous cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare overall survival (OS) in patients with advanced stage refractory squamous cell carcinoma (SCCA) of the lung randomized to nivolumab plus ipilimumab versus nivolumab.

SECONDARY OBJECTIVES:

I. To compare investigator-assessed progression-free survival (IA-PFS) in patients with advanced stage refractory SCCA of the lung randomized to nivolumab plus ipilimumab versus nivolumab.

II. To compare the response rates (confirmed and unconfirmed, complete and partial) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 among patients randomized to receive nivolumab plus ipilimumab versus nivolumab.

III. To compare the response rates (confirmed only, complete and partial) per RECIST 1.1 among patients randomized to receive nivolumab plus ipilimumab versus nivolumab.

IV. To evaluate the frequency and severity of toxicities associated with nivolumab plus ipilimumab versus nivolumab.

TRANSLATIONAL MEDICINE OBJECTIVES:

I. To evaluate if there is a differential treatment effect on OS, IA-PFS, and response by tumor programmed death-ligand 1 (PD-L1) expression status.

II. To examine patient reported outcomes by treatment arm.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 and ipilimumab IV over 60 minutes on day 1 of every third course (every 42 days). Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive nivolumab IV over 30 minutes on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment but prior to disease progression, patients are followed up every 3 months for 1 year and then every 6 months for up to 3 years. After disease progression, patients are followed up every 6 months for 2 years and at end of year 3 after sub-study registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all SCREENING/PRE-SCREENING and SUB-STUDY REGISTRATION COMMON ELIGIBILITY CRITERIA as specified in S1400: Phase II/III Biomarker-Driven Master Protocol for Previously Treated Squamous Cell Lung Cancer (Lung-Map)
* Patients must have been assigned to S1400I
* Patients must not have had prior treatment with an anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2, anti-cytotoxic T-lymphocyte-associated protein (CTLA)-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways
* Patients must not have an active, known, or suspected autoimmune disease; patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients must not have any known allergy or reaction to any component of the nivolumab and ipilimumab formulations
* Patients must not have received systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days prior to sub-study registration; inhaled or topical steroids, and adrenal replacement doses =< 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease
* Patients must not have a known positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection; patients with a positive hepatitis C antibody with a negative viral load are allowed
* Patients must not have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Patients must not have interstitial lung disease that is symptomatic or disease that may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Patients must also be offered participation in banking for future use of specimens
* Patients must have a lipase, amylase, TSH with reflex free T3/T4 performed within 7 days prior to sub-study registration
* Patients must not have any grade III/IV cardiac disease as defined by the New York Heart Association Criteria (i.e., patients with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), unstable angina pectoris, and myocardial infarction within 6 months, or serious uncontrolled cardiac arrhythmia

  * Patients with a history of congestive heart failure (CHF) or at risk because of underlying cardiovascular disease or exposure to cardiotoxic drug should have an electrocardiogram (EKG) and echocardiogram performed to evaluate cardiac function as clinically indicated
  * Patients with evidence of congestive heart failure (CHF), myocardial infarction (MI), cardiomyopathy, or myositis should have a cardiac evaluation including lab tests and cardiology consultations as clinically indicated including EKG, creatine phosphokinase (CPK), troponin, and echocardiogram
* Patients who can complete Patient Reported Outcomes (PRO) forms in English are required to complete a pre-study S1400I Patient Reported Outcomes (PRO) Questionnaire and a pre-study S1400I European Quality of Life Five Dimension (EQ-5D) Questionnaire within 14 days prior to registration; NOTE: Patients enrolled to S1400I prior to 9/1/2016 are not eligible for the PRO study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2026-04-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vassiliki Papadimitrakopoulou, Principal Investigator — SWOG Cancer Research Network
Locations (1207):
- United States (1201):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Yuma Cancer Center, Yuma, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - City of Hope Corona, Corona, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - City of Hope Mission Hills, Mission Hills, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - Pacific Cancer Care-Monterey, Monterey, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Feather River Cancer Center, Paradise, California
  - City of Hope Rancho Cucamonga, Rancho Cucamonga, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Northbay Cancer Center, Vacaville, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Yale-New Haven Shoreline Medical Center, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Midstate Medical Center, Meriden, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Lawrence and Memorial Cancer Center, Waterford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Hawaii Oncology Inc-POB I, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - AMITA Health Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - AMITA Health Cancer Institute and Outpatient Center, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - AMG Oncology - Naperville, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Deaconess Clinic Downtown, Evansville, Indiana
  - IU Health Central Indiana Cancer Centers-Fishers, Fishers, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Richard L. Roudebush Veterans Affairs Medical Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - The Community Hospital, Munster, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - JCHC McCreery Cancer Center, Fairfield, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - King's Daughter's Medical Center, Ashland, Kentucky
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Hardin Memorial Hospital, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Norton Audubon Hospital and Medical Campus, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Mary Bird Cancer Center/Saint Tammany Parish, Covington, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center/Terrebonne General Medical Center, Houma, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Robert Veith MD LLC, Metairie, Louisiana
  - University Health-Conway, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - LSU Healthcare Network/Saint Charles, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Waldo County General Hospital, Belfast, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Mercy Hospital, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Upper Chesapeake Medical Center, Bel Air, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Western Maryland Regional Medical Center, Cumberland, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Kensington Medical Center, Kensington, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - MedStar Montgomery Medical Center, Olney, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Veteran's Administration Medical Center - Ann Arbor, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute?Downriver, Brownstown, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Point, Grosse Pointe, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Lymphoma Clinic of Michigan, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Assarian Cancer Center, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon and Rectal Association, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Hematology Oncology Consultants PC, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Saint Joseph Health System-Tawas City, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Bhadresh Nayak MD PC-Warren, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - The University of Kansas Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Nevada Cancer Specialists-Saint Rose, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - Nevada Cancer Specialists?Oakey, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Nevada Cancer Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Specialists-Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Alpine Hematology-Oncology, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Reno Oncology Consultants, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Ocean Medical Center, Brick, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Bayshore Community Hospital, Holmdel, New Jersey
  - Southern Ocean County Medical Center, Manahawkin, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital-Luckow Pavilion, Paramus, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Neurosurgeons of New Jersey-Ridgewood, Ridgewood, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Lovelace Medical Center-Downtown, Albuquerque, New Mexico
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - New York Oncology Hematology PC -Albany Medical Center, Albany, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - Asheville Hematology-Oncology Associates, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Durham Veterans Affairs Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Health, Hendersonville, North Carolina
  - Hayworth Cancer Center, High Point, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Lake Norman Hematology Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Lake Norman Hematology Oncology Specialists-Mooresville, Mooresville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physicians LLC-Samaritan North, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Ireland Cancer Center Landerbrook Health Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Ireland Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University Pointe, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates-Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates PA-Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Boston Baskin Cancer Center-Bartlett, Bartlett, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Cancer Survival Center - West, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Family Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Thompson Oncology Group-Oak Ridge, Oak Ridge, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Texas Oncology at Baylor Charles A Sammons Cancer Center, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - MD Anderson Regional Care Center-Katy, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - University Medical Center, Lubbock, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - MD Anderson Regional Care Center-Bay Area, Nassau Bay, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson Regional Care Center-Sugar Land, Sugar Land, Texas
  - MD Anderson Regional Care Center-The Woodlands, The Woodlands, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont College of Medicine, Burlington, Vermont
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Seattle Cancer Care Alliance at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Spokane Valley Cancer Center-Mayfair, Spokane, Washington
  - Cancer Care Northwest-Valley, Spokane, Washington
  - Spokane Valley Cancer Center-Mission, Spokane, Washington
  - Cancer Care Northwest-North Spokane, Spokane, Washington
  - Rockwood North Cancer Treatment Center, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology SC-Appleton, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center - Eau Claire, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - The Alyce and Elmore Kraemer Cancer Care Center, West Bend, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Saint Clare's Hospital, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Lee SM, Fan W, Wang A, Vaidya R, Redman MW, Gettinger SN, Bazhenova L, Herbst RS, Hershman DL, Unger JM. Novel Approaches for Dynamic Visualization of Adverse Event Data in Oncology Clinical Trials: A Case Study Using Immunotherapy Trial S1400-I (SWOG). JCO Clin Cancer Inform. 2023 Apr;7:e2200165. doi: 10.1200/CCI.22.00165. PMID 37084329
- [Derived] Gettinger SN, Redman MW, Bazhenova L, Hirsch FR, Mack PC, Schwartz LH, Bradley JD, Stinchcombe TE, Leighl NB, Ramalingam SS, Tavernier SS, Yu H, Unger JM, Minichiello K, Highleyman L, Papadimitrakopoulou VA, Kelly K, Gandara DR, Herbst RS. Nivolumab Plus Ipilimumab vs Nivolumab for Previously Treated Patients With Stage IV Squamous Cell Lung Cancer: The Lung-MAP S1400I Phase 3 Randomized Clinical Trial. JAMA Oncol. 2021 Sep 1;7(9):1368-1377. doi: 10.1001/jamaoncol.2021.2209. PMID 34264316
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 275 enrolled patients, 252 were deemed eligible (125 randomized to nivolumab/ipilimumab and 127 to nivolumab).
Period: Overall Study
Arm/Group | Arm I (Nivolumab, Ipilimumab) | Arm II (Nivolumab)
Started | 125 | 127
Completed | 0 | 0
Not Completed | 125 | 127
Not completed — Adverse Event | 31 | 19
Not completed — Refusal unrelated to adverse events | 10 | 5
Not completed — Disease progression/relapse | 61 | 89
Not completed — Death | 11 | 7
Not completed — Other- not protocol specified | 6 | 4
Not completed — On protocol treatment | 6 | 3

BASELINE CHARACTERISTICS:
Population: Eligible and evaluable participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Nivolumab, Ipilimumab) | Arm II (Nivolumab) | Total
Number analyzed (Participants) | 125 | 127 | 252
Age, Continuous [Median (Full Range); unit: years] | 67.5 [41.8 to 83.4] | 68.1 [48.6 to 90.3] | 67.5 [41.8 to 90.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 41 | 83
  Male | 83 | 86 | 169
Race/Ethnicity, Customized [Number; unit: participants]
  White | 102 | 104 | 206
  Black | 17 | 16 | 33
  Asian | 0 | 4 | 4
  Pacific Islander | 0 | 1 | 1
  Native American | 1 | 2 | 3
  Multiracial | 1 | 0 | 1
  Unknown race | 4 | 0 | 4
  Hispanic ethnicity | 2 | 1 | 3
  Unknown ethnicity | 3 | 0 | 3
No. of prior systemic therapies for stage IV or recurrent disease [Count of Participants; unit: Participants] — The "0" category includes patients who received systemic therapy for stage I to III non-small cell lung cancer within 1 y of S1400I treatment.
  Participants
    0 | 35 | 35 | 70
    1 | 73 | 77 | 150
    2 | 6 | 7 | 13
    ≥3 | 3 | 1 | 4
    Unknown | 8 | 7 | 15
Zubrod performance score [Count of Participants; unit: Participants] — Participants were graded according to the Zubrod Performance Status Scale. 0 - Fully active, able to carry out on all pre-disease performance without restriction.
  1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light housework, office work.
  Participants
    0 | 36 | 35 | 71
    1 | 89 | 92 | 181
Weight loss in past 6 months [Count of Participants; unit: Participants]
  <5% | 86 | 93 | 179
  5% to <10% | 25 | 18 | 43
  10% to <20% | 13 | 13 | 26
  ≥20% | 1 | 3 | 4
Smoking status [Count of Participants; unit: Participants]
  Current | 48 | 54 | 102
  Former | 75 | 72 | 147
  Never | 2 | 1 | 3
Brain metastases at baseline [Count of Participants; unit: Participants] | 8 | 12 | 20
Liver metastases at baseline [Count of Participants; unit: Participants] | 23 | 30 | 53
Prior radiation therapy [Number; unit: participants]
  Localized radiation | 36 | 49 | 85
  Radiation with curative intent | 41 | 45 | 86

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Duration from randomization to death due to any cause
Time Frame: From date of registration to maximum of 3 years or death
Population: Eligible and evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Nivolumab, Ipilimumab) | Arm II (Nivolumab)
Number analyzed (Participants) | 125 | 127
months | 10 [8.0 to 14.4] | 11 [8.6 to 13.7]

2. Secondary Outcome: Investigator-assessed Progression-free Survival (IA-PFS)
Description: Duration from randomization to first occurrence of progression by RECIST 1.1, symptomatic deterioration, or death due to any cause. The IA-PFS for patients last known to be alive and free of progression or symptomatic deterioration was censored at the date of last disease assessment.
  Progression is defined as one or more of the following: 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline as well as an absolute increase of at least 0.5 cm; Unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided); Appearance of any new lesion/site; Death due to disease without prior documentation of progression and without symptomatic deterioration
Time Frame: From date of registration to maximum of 3 years or death
Population: Eligible and evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Nivolumab, Ipilimumab) | Arm II (Nivolumab)
Number analyzed (Participants) | 125 | 127
months | 3.8 [2.7 to 4.4] | 2.9 [1.8 to 4.0]

3. Secondary Outcome: Objective Response Rate
Description: Response was defined as the occurrence of a complete or partial response, confirmed or unconfirmed per RECIST 1.1 criteria. Response for patients not known to have a response was coded as nonresponse.
  Complete response: Complete disappearance of all target and non-target lesions. No new lesions. No disease related symptoms. Any lymph nodes (whether target or non-target) must have reduction in short axis to < 1.0 cm. All disease must be assessed using the same technique as baseline.
  Partial response: Applies only to patients with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. All target measurable lesions must be assessed using the same techniques as baseline.
Time Frame: From date of registration to maximum of 3 years or death
Population: Eligible and evaluable participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Nivolumab, Ipilimumab) | Arm II (Nivolumab)
Number analyzed (Participants) | 125 | 127
percentage of participants | 18 [12 to 25] | 17 [10 to 23]

4. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported. CTCAE Version 4.0 was used for routine toxicity reporting and CTCAE Version 5.0 was used for reporting SAEs.
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Population: Participants who received at least one dose of protocol treatment
Measure: Number; unit: Participants
Groups:
- Nivolumab + Ipilimumab: Participants receive nivolumab on day 1 of each 14-day cycle and ipilimumab on day 1 of every third cycle beginning with cycle 1.
  Nivolumab: Given IV Durvalumab: Given IV
- Nivolumab: Participants receive nivolumab on day 1 of each 14-day cycle.
  Nivolumab: Given IV.
Arm/Group | Nivolumab + Ipilimumab | Nivolumab
Number analyzed (Participants) | 124 | 123
Participants
  Abdominal pain | 1 | 0
  Acute kidney injury | 1 | 1
  Alanine aminotransferase increased | 5 | 2
  Alkaline phosphatase increased | 2 | 2
  Anemia | 5 | 1
  Anorexia | 2 | 2
  Arthralgia | 2 | 0
  Aspartate aminotransferase increased | 6 | 2
  Atrioventricular block complete | 1 | 0
  Autoimmune disorder | 1 | 0
  Blood bilirubin increased | 0 | 2
  Cardiac arrest | 1 | 0
  Cardiac troponin I increased | 1 | 0
  Chronic kidney disease | 0 | 1
  Colitis | 1 | 3
  Confusion | 2 | 0
  Constipation | 1 | 0
  Death NOS | 1 | 0
  Dehydration | 2 | 0
  Diarrhea | 3 | 2
  Dyspnea | 5 | 5
  Enterocolitis | 1 | 0
  Erythroderma | 1 | 0
  Fall | 1 | 0
  Fatigue | 11 | 7
  General disorders and admin site conditions - Other | 1 | 0
  Generalized muscle weakness | 3 | 1
  Headache | 0 | 1
  Heart failure | 1 | 0
  Hepatic failure | 1 | 0
  Hepatobiliary disorders - Other, specify | 1 | 0
  Hypercalcemia | 2 | 0
  Hyperglycemia | 1 | 1
  Hyperkalemia | 1 | 0
  Hypertension | 4 | 1
  Hyperthyroidism | 1 | 0
  Hypoalbuminemia | 2 | 0
  Hypokalemia | 3 | 3
  Hyponatremia | 7 | 3
  Hypotension | 2 | 0
  Hypoxia | 4 | 1
  Infections and infestations - Other, specify | 0 | 1
  Insomnia | 1 | 0
  Leukocytosis | 1 | 0
  Lipase increased | 6 | 1
  Lung infection | 2 | 6
  Lymphocyte count decreased | 3 | 5
  Memory impairment | 0 | 1
  Myalgia | 1 | 0
  Myocarditis | 1 | 0
  Myositis | 1 | 0
  Nausea | 0 | 2
  Pancreatitis | 0 | 1
  Periorbital edema | 1 | 0
  Pleural effusion | 1 | 0
  Pneumonitis | 9 | 6
  Proteinuria | 0 | 1
  Pruritus | 2 | 0
  Rash maculo-papular | 3 | 1
  Resp, thoracic and mediastinal disorders - Other | 2 | 1
  Respiratory failure | 2 | 0
  Sepsis | 1 | 1
  Serum amylase increased | 2 | 1
  Skin and subcutaneous tissue disorders - Other | 1 | 0
  Skin infection | 2 | 0
  Sore throat | 1 | 0
  Stroke | 1 | 0
  Supraventricular tachycardia | 1 | 0
  Syncope | 1 | 0
  Thromboembolic event | 1 | 1
  Treatment related secondary malignancy | 0 | 1
  Vomiting | 1 | 1
  Weight gain | 0 | 1
  Weight loss | 1 | 0

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Description: CTCAE Version 4.0 was used for routine toxicity reporting and CTCAE Version 5.0 was used for SAE reporting. All-Cause Mortality was assessed for all 252 eligible participants: 125 in the nivolumab/ipilimumab arm and 127 in the nivolumab arm. SAEs and other AEs were assessed for the 247 participants who received protocol therapy: 124 in the nivolumab/ipilimumab arm and 123 in the nivolumab arm.
Arm/Group | Nivolumab + Ipilimumab | Nivolumab
All-Cause Mortality (participants affected / at risk) | 92/125 | 105/127
Serious Adverse Events (participants affected / at risk) | 78/124 | 58/123
Other Adverse Events (participants affected / at risk) | 122/124 | 123/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab (N=124) | Nivolumab (N=123)
Anemia (Blood and lymphatic system disorders) | 8 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Heart failure (Cardiac disorders) | 3 | 1
Myocardial infarction (Cardiac disorders) | 5 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2
Pericardial tamponade (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 4 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Retinal vascular disorder (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0
Chills (General disorders) | 1 | 0
Death NOS (General disorders) | 6 | 4
Edema limbs (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 4
Fever (General disorders) | 4 | 2
Flu like symptoms (General disorders) | 2 | 0
Hypothermia (General disorders) | 1 | 0
Localized edema (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 2
Pain (General disorders) | 0 | 1
Sudden death NOS (General disorders) | 0 | 2
Hepatobiliary disorders-Other (Hepatobiliary disorders) | 1 | 2
Autoimmune disorder (Immune system disorders) | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1
Bronchial infection (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Infections and infestations-Other (Infections and infestations) | 2 | 1
Lung infection (Infections and infestations) | 13 | 10
Mucosal infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 5 | 3
Skin infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 2
Alkaline phosphatase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 3
Blood bilirubin increased (Investigations) | 1 | 1
Cardiac troponin I increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Lipase increased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 2 | 1
Serum amylase increased (Investigations) | 1 | 0
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 8 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 9
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 1
Dysphasia (Nervous system disorders) | 0 | 1
Edema cerebral (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Nervous system disorders-Other (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 2
Confusion (Psychiatric disorders) | 6 | 4
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Psychosis (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 7 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 | 13
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Erythroderma (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 4 | 3
Thromboembolic event (Vascular disorders) | 4 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab (N=124) | Nivolumab (N=123)
Anemia (Blood and lymphatic system disorders) | 58 | 48
Sinus tachycardia (Cardiac disorders) | 11 | 6
Hyperthyroidism (Endocrine disorders) | 14 | 10
Hypothyroidism (Endocrine disorders) | 23 | 18
Blurred vision (Eye disorders) | 9 | 5
Eye disorders-Other (Eye disorders) | 8 | 4
Abdominal pain (Gastrointestinal disorders) | 20 | 15
Constipation (Gastrointestinal disorders) | 34 | 29
Diarrhea (Gastrointestinal disorders) | 37 | 42
Dry mouth (Gastrointestinal disorders) | 18 | 7
Dysphagia (Gastrointestinal disorders) | 8 | 11
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 | 7
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 5 | 8
Mucositis oral (Gastrointestinal disorders) | 7 | 6
Nausea (Gastrointestinal disorders) | 45 | 44
Vomiting (Gastrointestinal disorders) | 22 | 25
Chills (General disorders) | 16 | 14
Edema limbs (General disorders) | 16 | 18
Fatigue (General disorders) | 69 | 75
Fever (General disorders) | 7 | 16
Flu like symptoms (General disorders) | 1 | 8
Non-cardiac chest pain (General disorders) | 8 | 18
Pain (General disorders) | 23 | 32
Infections and infestations-Other (Infections and infestations) | 6 | 7
Lung infection (Infections and infestations) | 8 | 13
Sinusitis (Infections and infestations) | 4 | 9
Skin infection (Infections and infestations) | 4 | 7
Upper respiratory infection (Infections and infestations) | 11 | 12
Urinary tract infection (Infections and infestations) | 3 | 7
Fall (Injury, poisoning and procedural complications) | 8 | 12
Alanine aminotransferase increased (Investigations) | 25 | 10
Alkaline phosphatase increased (Investigations) | 29 | 25
Aspartate aminotransferase increased (Investigations) | 22 | 13
Blood bilirubin increased (Investigations) | 9 | 7
Creatinine increased (Investigations) | 19 | 17
Investigations-Other (Investigations) | 19 | 20
Lipase increased (Investigations) | 11 | 11
Lymphocyte count decreased (Investigations) | 27 | 25
Platelet count decreased (Investigations) | 21 | 8
Serum amylase increased (Investigations) | 10 | 8
Weight loss (Investigations) | 34 | 27
White blood cell decreased (Investigations) | 8 | 4
Anorexia (Metabolism and nutrition disorders) | 48 | 45
Dehydration (Metabolism and nutrition disorders) | 13 | 13
Hypercalcemia (Metabolism and nutrition disorders) | 12 | 12
Hyperglycemia (Metabolism and nutrition disorders) | 25 | 32
Hyperkalemia (Metabolism and nutrition disorders) | 9 | 14
Hypoalbuminemia (Metabolism and nutrition disorders) | 48 | 48
Hypocalcemia (Metabolism and nutrition disorders) | 15 | 16
Hypoglycemia (Metabolism and nutrition disorders) | 7 | 7
Hypokalemia (Metabolism and nutrition disorders) | 35 | 21
Hypomagnesemia (Metabolism and nutrition disorders) | 37 | 26
Hyponatremia (Metabolism and nutrition disorders) | 46 | 43
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 12 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 15
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 15
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 19 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 21
Dizziness (Nervous system disorders) | 21 | 21
Dysgeusia (Nervous system disorders) | 5 | 10
Headache (Nervous system disorders) | 16 | 19
Peripheral sensory neuropathy (Nervous system disorders) | 11 | 13
Anxiety (Psychiatric disorders) | 15 | 15
Confusion (Psychiatric disorders) | 9 | 6
Depression (Psychiatric disorders) | 6 | 10
Insomnia (Psychiatric disorders) | 12 | 20
Hematuria (Renal and urinary disorders) | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 43 | 42
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 46 | 58
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 | 14
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Wheezing (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 31 | 24
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 31 | 18
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 12 | 9
Hot flashes (Vascular disorders) | 0 | 7
Hypertension (Vascular disorders) | 19 | 12
Hypotension (Vascular disorders) | 14 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT02785952/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT02785952/ICF_001.pdf